CLINICAL TRIAL: NCT00871013
Title: UARK 2008-03 Phase II Trial for Patients Not Qualifying for TT4 and TT5 Protocols Because of Prior Therapy (No Prior Transplant)
Brief Title: Trial for Patients Not Qualifying for TT4 and TT5 Protocols Because of Prior Therapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 108053
Record Dates: First submitted 2009-03-27; First posted 2009-03-30 (Estimated); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Myeloma
Keywords: improve remission rate & survival time in high-risk myeloma
MeSH Terms: conditions — Neoplasms, Plasma Cell | interventions — Melphalan; Bortezomib; Thalidomide; Dexamethasone; Calcium Dobesilate; Cisplatin; Doxorubicin; Cyclophosphamide; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MEL-VTD-PACE (Experimental): Melphalan, Velcade, Thalidomide, Dexamethasone, CisPlatin, Adriamycin, Cyclophosphamide, Etoposide
  Interventions: Drug: Melphalan; Drug: Velcade; Drug: Thalidomide; Drug: Dexamethasone; Drug: Cisplatin; Drug: Adriamycin; Drug: Cyclophosphamide; Drug: Etoposide

INTERVENTIONS:
Drug: Melphalan — Given by vein, Day 3
  First Inter-Therapy Treatment Bortezomib (Velcade) By vein Days 1 and 4
  Second Inter-Therapy Treatment Bortezomib (Velcade) By vein Days 1 and 4
  Second Transplant Bortezomib (Velcade) By vein Day -5 and Day -2
  Year 1 Maintenance Velcade (bortezomib) By vein Days 1, 8, 15, 22(weekly) Every 28 days
  Years 2 & 3 Maintenance Velcade (bortezomib) By vein Days 1, 8, 15, 22(weekly) Every 56 days
  Other Names: Alkeran
Drug: Velcade — Given by vein, Days 1, 5, 8, 11
  Other Names: Bortezomib, PS-341
Drug: Thalidomide — Given by mouth at bedtime, Days 5-8
  Other Names: Thalomid
Drug: Dexamethasone — Given by mouth, once per day Days 5-8
  Other Names: Decadron
Drug: Cisplatin — Given by vein, Days 5-8 continuous infusion
  Other Names: Platinol, CDDP
Drug: Adriamycin — Given by vein, days 5-8 continuous infusion
  Other Names: Doxorubicin
Drug: Cyclophosphamide — Given by vein days 5-8 continuous infusion
  Other Names: Cytoxan
Drug: Etoposide — Given by vein days 5-8 continuous infusion
  Other Names: Vepesid, VP-16

SUMMARY:
There have been four previous Total Therapy (TT1 through IIIB) studies for multiple myeloma at the MIRT from 1989 to present. Results have shown that participants treated on these studies had better outcomes (meaning they have lived longer and had better responses to treatment) when compared to individuals treated with standard chemotherapy.

Past studies conducted at the MIRT have shown that participants presenting to MIRT who have already received treatment for myeloma tend to have shorter remissions (disappearance of signs and symptoms of myeloma) and do not survive as long as participants who come to MIRT with untreated myeloma. Researchers at MIRT think that one reason for this is may be that the myeloma cells re-grow in the time when participants are not receiving treatment because they are recovering from high-dose chemotherapy. In this study, participants will receive several chemotherapy drugs previously shown to be effective in myeloma, but in lower doses and in shorter cycles. It is hoped that by giving the drugs in this way, myeloma cells will not have time to re-grow between cycles, therefore resulting in longer remissions. This study is being done in an attempt to improve the remission rate and the survival time for participants with high-risk myeloma.

DETAILED DESCRIPTION:
* To find out if giving multi-agent chemotherapy in lower and more frequent doses to make the timely delivery of chemotherapy cycles possible, will result in better myeloma responses
* To find out if changing the way the drugs are given during the transplant phase will also result in fewer side effects, while still being effective
* To find out if giving treatment between transplants (called "inter-therapy") will prevent the myeloma from re-growing between transplants
* To find out if long-term maintenance therapy will result in longer remissions
* To find out what the effects (good and bad) of this overall treatment will be
* To learn more about the biology and genetics of multiple myeloma by performing imaging tests and collecting blood, bone marrow aspirate and biopsies, and biopsies of lesions seen on MRI or PET scans. Bone marrow aspirates and biopsies are tissue sample collected from the bone cavity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic multiple myeloma (MM), with at least one prior line of chemotherapy or newly diagnosed without any prior therapy.
* Zebroid ≤ 2, unless solely due to symptoms of MM-related bone disease (Appendix 4).
* Patients must be at least 18 years of age and not older than 75 years of age at the time of registration.
* Patient must not have had a prior auto- or allotransplant.
* Patient must have signed an IRB-approved informed consent and understand the investigational nature of the study.
* Patients must have adequate pulmonary function studies ≥ 50% of predicted on mechanical aspects (FEV1, FVC, etc) and diffusion capacity (DLCO) ≥ 50% of predicted, within 60 days prior to enrollment. Patients unable to complete pulmonary function tests because of myeloma-related chest pain, must have a high resolution CT scan of the chest and must also have acceptable arterial blood gases defined as P02 greater than 70.
* Ejection fraction by ECHO or MUGA must be ≥ 40% and must be performed within 60 days prior to enrollment, unless the patient has received chemotherapy within that period of time (dexamethasone and thalidomide excluded), in which case the LVEF must be repeated.
* Patients must not have prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has not received treatment for one year prior to enrollment. Other cancers will only be acceptable if the patient's life expectancy exceeds five years.
* Patients must be able to receive full doses of Mel-VRD-PACE, in the opinion of the treating investigator, with the exception that patients with creatinine clearance 30-50 ml/min will receive only 50% of the cisplatin dose.

Exclusion Criteria:

* Fever or active infection requiring intravenous antibiotic, defined as fever or antibiotics within 72 hours from registration.
* Severe renal dysfunction, defined as a creatinine > 3mg/dl or a creatinine clearance of < 30ml/min.
* Significant neurotoxicity, defined as grade ≥ 3 neurotoxicity per NCI Common Toxicity Criteria (See Appendix).
* Platelet count < 30,000/mm3, and ANC < 1,000/μl
* POEMS Syndrome: (Polyneuropathy, Organomegaly, Endocrinopathy, Monoclonal gammopathy, and Skin changes
* Clinically significant hepatic dysfunction as noted by direct bilirubin or AST >3 times the upper normal limit or clinically significant concurrent hepatitis.
* New York Heart Association (NYHA) Class III or Class IV heart failure (Appendix 4).
* Recent (≤ 6 months) myocardial infarction, unstable angina, difficult to control congestive heart failure, uncontrolled hypertension, or difficult to control cardiac arrhythmias are ineligible.
* Patients with a history of treatment for clinically significant ventricular cardiac arrhythmias.
* Poorly-controlled hypertension, diabetes mellitus, or other serious medical illness or psychiatric illness that could potentially interfere with the completion of treatment according to this protocol.
* Prior cumulative total of Adriamycin exposure >450 mg/m2.
* Prior exposure to thalidomide which resulted in severe toxicity requiring drug discontinuation.
* Prior exposure to Revlimid which resulted in severe toxicity requiring drug discontinuation
* Hypersensitivity to boron, or Mannitol. Prior exposure to bortezomib which resulted in severe toxicity requiring drug discontinuation.
* Pregnant or nursing women may not participate. Women of childbearing potential must have a negative pregnancy documented within one week of registration. Women/men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2009-03; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is to assess the continued complete and near complete response rate (CR/nCR) at two years after initiation of therapy. . | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Zangari, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Davies FE, Rosenthal A, Rasche L, Petty NM, McDonald JE, Ntambi JA, Steward DM, Panozzo SB, van Rhee F, Zangari M, Schinke CD, Thanendrarajan S, Walker B, Weinhold N, Barlogie B, Hoering A, Morgan GJ. Treatment to suppression of focal lesions on positron emission tomography-computed tomography is a therapeutic goal in newly diagnosed multiple myeloma. Haematologica. 2018 Jun;103(6):1047-1053. doi: 10.3324/haematol.2017.177139. Epub 2018 Mar 22. PMID 29567784
- See also: Multiple Myeloma — http://myeloma.uams.edu/